CLINICAL TRIAL: NCT06661343
Title: A Multi-Level Integrated Strategy to Optimize PrEP Adherence for Black MSM and Accelerate Implementation at Scale
Brief Title: Pre-exposure Prophylaxis (PrEP) Adherence for Black MSM
Acronym: C4+3MV
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 2000037790; 1R01MH138225-01 (NIH)
Record Dates: First submitted 2024-10-24; First posted 2024-10-28 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: HIV Prevention; PrEP Adherence; HIV Risk Reduction
Keywords: HIV; PrEP; Black MSM; Adherence; HIV Prevention; Stigma Reduction; C4 Intervention; 3MV Program; Behavioral Health

STUDY DESIGN:
Intervention Model Description: This study uses a stepped-wedge cluster randomized trial. Participants from multiple networks are introduced to the intervention in a sequential manner, with each cluster beginning in a control phase and transitioning into one of two intervention phases over time. This design allows for comparison between groups while also ensuring all participants eventually receive the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- C4 Intervention (Experimental): Participants in this arm will receive care coordination and support through the C4 intervention. This program focuses on addressing structural barriers, such as healthcare access and mental health, to improve PrEP adherence. Participants will also attend regular counseling sessions and have their PrEP use monitored through dried blood spot (DBS) tests.
  Interventions: Behavioral: C4 Program
- C4 + 3MV Intervention (Experimental): Participants in this arm will receive the C4 intervention, along with the 3MV (Many Men, Many Voices) behavioral intervention. The 3MV program aims to reduce stigma, promote safer behaviors, and increase self-efficacy. This arm integrates both structural and behavioral approaches to enhance PrEP adherence. Participants will complete counseling sessions, group activities, and DBS testing for monitoring adherence.
  Interventions: Behavioral: C4 + 3MV Program

INTERVENTIONS:
Behavioral: C4 Program — The C4 intervention is a behavioral program designed to provide care coordination to address structural barriers to PrEP adherence among Black men who have sex with men (MSM). It includes personalized support services, focusing on healthcare access, mental health, and stigma reduction to promote consistent PrEP use. Participants will receive counseling sessions and follow-ups based on their individual needs.
  Other Names: Client Centered Care Coordination
  Arms: C4 Intervention
Behavioral: C4 + 3MV Program — This intervention combines the C4 care coordination with the 3MV behavioral program. The 3MV program focuses on behavior change, addressing self-efficacy, stigma, and promoting healthy practices. Through this combination, participants receive both structural and behavioral support to maximize their adherence to PrEP.
  Other Names: Many Men Many Voices and Client Centered Care Coordination Integrated Intervention
  Arms: C4 + 3MV Intervention

SUMMARY:
The goal of this clinical trial is to learn if two interventions-C4 and C4+3MV-can improve PrEP adherence (taking medication to prevent HIV) among Black men who have sex with men (MSM). The study will also explore the most effective ways to support participants in continuing their PrEP use over time.

The main questions it aims to answer are:

* Does the C4 program help participants take PrEP more regularly?
* Does adding the 3MV intervention to C4 provide additional support for adherence?

Researchers will compare two intervention strategies to see if they result in better PrEP adherence:

* C4 Intervention: A program focused on individualized care coordination and addressing structural needs.
* C4 + 3MV Intervention: A combination of care coordination with additional behavioral change sessions.

Participants will:

* Participate in PrEP education and counseling sessions.
* Have their PrEP use monitored through dried blood spot (DBS) tests.
* Complete questionnaires about their experiences and challenges with PrEP. Receive support sessions tailored to address individual barriers to PrEP adherence.

DETAILED DESCRIPTION:
This clinical trial aims to evaluate two intervention strategies-C4 and C4 + 3MV-to improve adherence to PrEP (pre-exposure prophylaxis) among Black men who have sex with men (MSM) in two metropolitan areas: Dallas/Fort Worth and Miami/Fort Lauderdale. The study addresses structural and behavioral barriers to PrEP adherence, aiming to reduce disparities in HIV prevention efforts.

Study Design and Methodology:

* Trial Type: Multi-site, staircase stepped-wedge randomized controlled trial (RCT)
* Duration: 24 months total, with 9-month intervention periods for each group
* Participants: 500 participants (250 at each site); Participants are recruited from community-based organizations and through network-based referrals

Randomization:

* 48 networks will be randomized into 8 sequences.
* Each network will experience a 3-month control period, followed by either the C4 intervention or the C4 + 3MV intervention.

Interventions:

* C4 Intervention: Focuses on care coordination, addressing participants' needs related to healthcare access, stigma, and mental health services. Uses individualized care plans and support systems to facilitate adherence.
* C4 + 3MV Intervention: Incorporates both care coordination and the 3MV (Many Men, Many Voices) behavioral change program. 3MV focuses on reducing stigma, promoting safe behaviors, and improving self-efficacy through group sessions.

Primary and Secondary Outcomes:

* Primary Outcome: PrEP adherence, measured through dried blood spot (DBS) assays to assess drug levels over time.
* Secondary Outcomes: Changes in HIV-related health-seeking behavior (e.g., frequency of HIV testing); Autonomy and social support, measured through validated scales; Reduction in stigma and mental health improvements

Data Collection and Monitoring:

* Data will be collected at multiple points using questionnaires, DBS tests, and counseling session evaluations.
* A Learn-as-You-Go (LAGO) adaptive analysis will be conducted every 6 months to optimize intervention delivery.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as male.
* Self-Identify as Black people.
* Aged 18 or older.
* Self Report having sex with men in the past 6 months.
* Eligible for PrEP or currently prescribed PrEP.
* Willing to participate in behavioral intervention sessions.

Exclusion Criteria:

* Currently diagnosed with HIV.
* Unable to provide informed consent.
* Unable to fully engage with the intervention due to health issues.
* Participating in another clinical trial with conflicting outcomes.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
PrEP adherence- self report | 0, 3, 6, 9, 12 months
  PrEP adherence will be assessed through self-report. Self-reported adherence is measured by doses taken in the past 30 days, with fewer missed doses indicating higher adherence.
PrEP adherence- biomarker validation | 0, 6, and 12 months
  PrEP adherence will be assessed through biomarker validation using dried blood samples. A tenofovir disoproxil fumarate (TFV-DF) level >700 fmol/punch confirms adherence.

SECONDARY OUTCOMES:
HIV Testing Frequency | Every 3 months for 12 months
  HIV testing frequency will be assessed by the number of tests taken in the past 90 days, with more tests indicating higher engagement in testing

OTHER OUTCOMES:
Perceived Competence for PrEP use | Baseline, 6 months, and 12 months
  Perceived Competence for PrEP Use Scale will measure participants' confidence in their ability to follow PrEP recommendations. Scores range from 9 to 45, with higher scores reflecting greater competence.
PrEP Use Self-Regulation | Baseline, 6 months, and 12 months
  PrEP Use Self-Regulation Questionnaire will assess participants' internalization of autonomous motivation to maintain adherence to PrEP. Scores range from 9 to 45, with higher scores indicating stronger self-regulation.
Basic Needs Satisfaction Scale | Every 3 months for 12 months
  The Basic Needs Satisfaction Scale (9 items) assesses participants' fulfillment of psychological needs (autonomy, competence, and relatedness) within social relationships, especially from close friends. Scores range from 9 to 45, with higher scores indicating greater satisfaction.
Healthcare Climate Questionnaire | Baseline, 6, and 12 months
  The Healthcare Climate Questionnaire (15 items) will measure participants' perception of their healthcare providers' support. Scores range from 15 to 75, with higher scores reflecting a more supportive healthcare environment.
Depression (PHQ-9) | Baseline, 6 months, and 12 months
  Depression will be assessed using the PHQ-9. PHQ-9 is a 9-item validated questionnaire used to screen for depression with a range of scores from 0-27. A cumulative score of ≥10 is considered positive with lower scores indicating no or mild anxiety.
HIV Stigma Scale | Baseline, 3, 6, 9, and 12 months
  Intersectional stigma will be measured across four subscales:
  Enacted Stigma (10 items) Vicarious Stigma (10 items) Perceived Stigma (10 items) Internalized Stigma (10 items) Each subscale ranges from 10 to 50, with higher scores indicating more stigma experienced.
Quality Client Perception of Coordination Quality | Baseline, 6 months, and 12 months
  The Client Perception of Coordination Quality Questionnaire will assess participants' satisfaction with healthcare services. Scores range from 3 to 15, with higher scores indicating better care coordination.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - South Florida Afro Pride Federation, Lauderdale Lakes, Florida
  - Abounding Prosperity, Inc., Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Investigators plan to share de-identified participant data, including information on PrEP usage, behavioral intervention participation, survey responses, and biological specimen results (e.g., dried blood spot test results). The shared data will support future research on HIV prevention and PrEP adherence, ensuring participant privacy throughout the process.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be made available within six months after the publication of the primary study results and will remain accessible for at least five years. The availability period may be extended depending on research needs and ethical guidelines.
Access Criteria: Access to the data will be granted to researchers with ethical approval from the Institutional Review Board (IRB). Researchers must submit a request outlining the purpose and intended use of the data, which will be reviewed by the study team. Approved users will be required to sign a Data Use Agreement to ensure the data is used for approved purposes only and that participant privacy is safeguarded.